CLINICAL TRIAL: NCT00400361
Title: A Dose-escalation Study of R1507 in Patients With Advanced Solid Tumors.
Brief Title: A Multiple Ascending Dose Study of R1507 in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO19373
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — RG-1507 monoclonal antibody

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RG1507

INTERVENTIONS:
Drug: RG1507 — Administered iv, either weekly or 3 weekly, at escalating doses (with a starting dose of 1mg/kg) (7 cohorts).

SUMMARY:
This study will determine the maximum tolerated dose and pharmacokinetic profile of R1507 in patients with metastatic or locally advanced malignant solid tumors, non-Hodgkin's lymphoma or Hodgkin's lymphoma. Groups of patients will be sequentially enrolled to receive ascending doses of R1507 either weekly or three-weekly by intravenous infusion. The starting dose of 1mg/kg iv for each dosing regimen will be escalated in subsequent groups of patients after a satisfactory assessment of safety, tolerability and pharmacokinetics of the previous dose. The anticipated time on study treatment is until disease progression or dose-limiting toxicity, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* solid neoplasm, non-Hodgkin's lymphoma or Hodgkin's lymphoma;
* metastatic or locally advanced disease, not curable by any currently available treatment.

Exclusion Criteria:

* severe, uncontrolled systemic disease;
* patients who require treatment with glucocorticoids or immunosuppressive treatment within last 6 months;
* patients with diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters, Cmax, Tmax, AUC, clearance, Vdss elimination half life | Throughout study

SECONDARY OUTCOMES:
Tumor response | Event driven

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Aurora, Colorado
  - New Brunswick, New Jersey
  - Houston, Texas

REFERENCES:
- [Derived] Xin Y, Xu F, Gao Y, Bhatt N, Chamberlain J, Sile S, Hammel S, Holt RJ, Ramanathan S. Pharmacokinetics and Exposure-Response Relationship of Teprotumumab, an Insulin-Like Growth Factor-1 Receptor-Blocking Antibody, in Thyroid Eye Disease. Clin Pharmacokinet. 2021 Aug;60(8):1029-1040. doi: 10.1007/s40262-021-01003-3. Epub 2021 Mar 26. PMID 33768488